CLINICAL TRIAL: NCT02801344
Title: The Impact of Protein Intake on Amino Acid and Protein Metabolism, and Performance During Intensified Training
Brief Title: The Impact of Protein Intake on Protein Metabolism During Intensified Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Moore, Associate professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PFE
Record Dates: First submitted 2016-05-25; First posted 2016-06-15 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: exercise; performance; recovery; muscle; protein
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal protein intake (Experimental): participants will receive the controlled-diet containing 0.8 g protein /kg/day and the test drink containing 0.14 g protein/kg/d.
  Interventions: Dietary Supplement: Normal; Other: Controlled-diet
- Moderate protein intake (Experimental): participants will receive the controlled-diet containing 1.20 g protein /kg/day and the test drink containing 0.40 g protein/kg/d.
  Interventions: Dietary Supplement: Moderate; Other: Controlled-diet
- High protein intake (Experimental): participants will receive the controlled-diet containing 1.83 g protein /kg/day and the test drink containing 1.03 g protein/kg/d.
  Interventions: Dietary Supplement: High; Other: Controlled-diet

INTERVENTIONS:
Dietary Supplement: Normal — test drink which contains low amount of amino acids (0.14 g/kg/day)
  Arms: Normal protein intake
Dietary Supplement: Moderate — test drink which contains moderate amount of amino acids (0.40 g/kg/day)
  Arms: Moderate protein intake
Dietary Supplement: High — test drink which contains high amount of amino acids (1.03 g/kg/day)
  Arms: High protein intake
Other: Controlled-diet — the diet containing 0.8 g protein /kg/day

SUMMARY:
Protein requirements in individuals who participate in endurance-based exercise training have been suggested to be greater than the current recommended dietary allowance (RDA).

Our recent study using the minimally invasive indicator amino acid oxidation (IAAO) technique have suggested that protein requirements in young men are at least 30% higher than the recommended protein intake.

The present study will investigate the impact of protein sufficiency on protein metabolism and performance during intensified training periods as a means to further our understanding of the nutritional requirements for the endurance athlete.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male, endurance-trained participants who have run regularly more than 45 km or 4.5 hours/week
* Participants who are categorized at least "very good" based on a study by Shvartz & Reibold [40], in which peak rate of oxygen consumption(VO2 Peak) is used as an index. (i.e. the participants whose VO2peak is ≥57 ml/kg/min (18-24 y), ≥54 ml/kg/min (25-29 y), ≥52 ml/kg/min (30-34 y), ≥49 ml/kg/min (35-39 y), ≥47 ml/kg/min (40-44 y), ≥44 ml/kg/min (45-50 y) according to his age,
* Participants who can cover 10 km in less than 60 min after the VO2peak test and 5 km Time trial on session 2.
* Participants will be 18-50 years old.
* Participants are willing to abide by the compliance rules of this study

Exclusion Criteria:

* Inability to meet health and physical activity guidelines according to the The Physical Activity Readiness Questionnaire for everyone.
* Female
* Inability to adhere to any of the compliance rules judged by principal investigator or medical doctor
* Regular tobacco use
* Illicit drug use (e.g. growth hormone, testosterone, etc.)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05; Primary Completion 2017-09 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change in 24h whole body protein balance | Difference between day 1 and day 4 whole body protein balance
  Protein balance (mg/kg/d; protein synthesis - protein breakdown) will be measured using [15N]Glycine method on day 1 and day 4 to determine the change over the intensified training period to compare between protein levels

SECONDARY OUTCOMES:
Change from baseline physical performance (5 km time trial) 5days after the beginning of training | 5days after the beginning of training
  Before and after 4 days of intensified training period, Duration (seconds) for completing 5-km running on treadmill will be measured.
change from baseline Physical performance (muscle strength) 5days after the beginning of training | 5days after the beginning of training
  Maximal strength will be assessed by a maximal isometric voluntary contraction (MVC), which will be tested for the knee-extensors using a custom-made knee-extension apparatus after 4 days intensified training.
change from baseline Physical Performance (muscle power) 5days after the beginning of training | 5days after the beginning of training
  Peak lower body power will be measured by force platform after 4days-intensified training.

OTHER OUTCOMES:
Creatine Phosphate Kinase activity on day 5 | 5days after the beginning of training
  Muscle damage markers (blood Creatine Phosphate Kinase activity, IU/L) will be compared between the experimental arms 5days after the beginning of training
Myoglobin concentration on day 5 | 5days after the beginning of training
  Muscle damage markers (blood Mb Concentration, mg/mL) will be compared between the experimental arms 5days after the beginning of training
IL-6 concentration on day 5 | 5days after the beginning of training
  inflammatory markers (IL-6 concentration, pg/ml) will be compared between the experimental arms 5days after the beginning of training
CRP concentration on day 5 | 5days after the beginning of training
  inflammatory markers (CRP concentration, mg/L) will be compared between the experimental arms 5days after the beginning of training
amino acid concentration on day 5 | 5days after the beginning of training
  amino acid concentration (mmol/mL) will be compared between the experimental arms 5days after the beginning of training

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Moore, Ph.D., Principal Investigator — Faculty of Kinesiology and Physical Education, University of Toronto
Locations (1):
- Goldring Centre For High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williamson E, Kato H, Volterman KA, Suzuki K, Moore DR. Greater plasma essential amino acids and lower 3-methylhistidine with higher protein intake during endurance training: a randomised control trial. Amino Acids. 2023 Oct;55(10):1285-1291. doi: 10.1007/s00726-022-03210-z. Epub 2022 Dec 7. PMID 36477889